CLINICAL TRIAL: NCT05817266
Title: Role of Field-Cycling Imaging in the Detection of Proctosigmoiditis Caused by Inflammatory Bowel Disease
Brief Title: Role of FCI in the Detection of Proctosigmoiditis Caused by IBD
Acronym: ROOFTOPS-IBD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding period ended
Sponsor: NHS Grampian (Other Government)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-093-22
Record Dates: First submitted 2023-03-10; First posted 2023-04-18 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases; Proctosigmoiditis
Keywords: Field-Cycling Imaging (FCI); Proctosigmoiditis; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Proctocolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proctosigmoiditis (Experimental): Participants with confirmed proctosigmoiditis will undergo one FCI scan.
  Interventions: Device: Field-cycling imaging (FCI)

INTERVENTIONS:
Device: Field-cycling imaging (FCI) — FCI scan

SUMMARY:
The goal of this pilot study is to explore the ability of field-cycling imaging, a new scanning technology being developed at the University of Aberdeen, to detect active disease in patients with proctosigmoiditis caused by inflammatory bowel disease.

DETAILED DESCRIPTION:
Field-cycling imaging (FCI) is an emerging technology that is being developed at the University of Aberdeen. It combines the use of a moderately high magnetic field (200mT) with the ability to probe low magnetic fields (0.2mT) so that image resolution can be preserved while also exploiting the high contrast present at low magnetic fields. This non-invasively provides quantitative data on the molecular dynamics in the tissues.

FCI represents a potentially new, non-invasive, way of assessing the extent and activity of inflammatory bowel disease (IBD). IBD can affect the rectum and distal sigmoid colon, this condition is called Proctosigmoiditis (PS). Currently, diagnosis of IBD depends on endoscopy for direct visualisation of the upper and lower gut, using CT scanning, with its attendant use of ionising radiation, and conventional MRI, particularly for the small bowel. Determining the activity of IBD remains a continuing challenge.

In this proof-of-concept study, the investigators will explore the ability of FCI to detect active disease in patients with PS.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of proctosigmoiditis, on the basis of a compatible history and previous flexible sigmoidoscopy
* Participants who are already under follow up in the NHS Grampian IBD clinic
* Participants must be between 16 and 80 years old
* Participants who meet the safety criteria for undergoing an MRI scan
* Participants who are able to fit inside the scanner
* Participants must be able to give fully informed consent
* Participants must be mobile enough to be positioned onto the FCI scanner couch

Exclusion Criteria:

* MRI-incompatible conditions, as detected in the MRI safety screening sheet
* Participants under 16 years old
* Participants who are unable to communicate in English
* Participants who are unable to give fully informed consent
* Women who are pregnant
* Restrictions to mobility that would prevent the correct positioning in the scanner
* Previous major abdominal surgery
* Any known significant comorbid disease that might interfere with treatment
* Malignancy or other conditions that would significantly reduce life expectancy
* Participants who suffer from claustrophobia

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Detection of proctosigmoiditis assessed by field-cycling imaging (FCI) scan | At baseline
  Validation of FCI T1 dispersion profiles as non-invasive technology able to detect proctosigmoiditis in participants with inflammatory bowel disease (IBD).

SECONDARY OUTCOMES:
Extent of proctosigmoiditis measured by field-cycling imaging (FCI) scan | At baseline
  Validation of FCI T1 dispersion profiles as a clinical tool for defining the extent of proctosigmoiditis in participants with inflammatory bowel disease (IBD).

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Bain, Dr, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No